CLINICAL TRIAL: NCT00130078
Title: Randomized Controlled Trial of SAVVY and HIV in Nigeria
Brief Title: Trial of SAVVY Vaginal Gel and HIV in Nigeria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosyn (Industry)
Collaborators: FHI 360 (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9784
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2005-09-26 (Estimated); Status verified 2005-08

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV transmission
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: 1.0% C31G SAVVY vaginal gel

SUMMARY:
Heterosexual contact is now the primary route of transmission for HIV worldwide. This study is a phase 3 trial designed to determine the effectiveness and safety of the 1.0% C31G (SAVVY) vaginal gel for the prevention of male-to-female transmission of HIV among women at high risk.

DETAILED DESCRIPTION:
Heterosexual contact is now the primary route of transmission for HIV worldwide. This study is a phase 3 multi-center, fully-masked, randomized, placebo controlled trial designed to determine the effectiveness and safety of the 1.0% C31G (SAVVY) vaginal gel for the prevention of male-to-female transmission of HIV among women at high risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 year old women
* HIV negative
* More than one sexual partner in past 3 months
* Average 3 coital acts per week
* Willing to use vaginal gel and condoms for 12 months

Exclusion Criteria:

* HIV positive
* Pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2142
Dates: Start 2004-09

PRIMARY OUTCOMES:
Combined incidence of HIV-1 and HIV-2

CONTACTS AND LOCATIONS:
Overall Officials: Paul Feldblum, Study Chair — FHI 360
Locations (2):
- Nigeria (2):
  - Department of Medical Microbiology & Parasitology, College of Medicine, University of Ibadan, Ibadan
  - Nigerian Institute of Medical Research, Lagos

REFERENCES:
- [Derived] Feldblum PJ, Adeiga A, Bakare R, Wevill S, Lendvay A, Obadaki F, Olayemi MO, Wang L, Nanda K, Rountree W. SAVVY vaginal gel (C31G) for prevention of HIV infection: a randomized controlled trial in Nigeria. PLoS One. 2008 Jan 23;3(1):e1474. doi: 10.1371/journal.pone.0001474. PMID 18213382